CLINICAL TRIAL: NCT01659281
Title: Efficacy of Artesunate-Mefloquine Combination Therapy for the Treatment of Uncomplicated Falciparum Malaria in Trat Province, Thailand
Brief Title: Efficacy of Artesunate-Mefloquine Combination Therapy in Trat Province, Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Responsible Party: Principal Investigator, Douglas Walsh, Dept Chief, Armed Forces Research Institute of Medical Sciences, Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR-1327
Record Dates: First submitted 2011-01-26; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Artesunate; Mefloquine; Plasmodium Falciparum; Thailand; Uncomplicated Plasmodium Falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 2-day oral treatment with: Artesunate 6mg/kg at 0 and 24 hours Mefloquine 25 mg/kg total dose split into 2 doses of 15 mg/kg at 0 hours and and 10 mg/kg given 6-24 hours later Primaquine 0.5 mg/kg single dose at 24 hours
  Interventions: Drug: Artesunate; Drug: Mefloquine
- 2 (Active Comparator): 3 days oral treatment with: Artesunate 4 mg/kg/day for 3 days Mefloquine 8 mg/kg/day for 3 days Primaquine 0.5 mg/kg single dose at 24 hours
  Interventions: Drug: Artesunate; Drug: Mefloquine

INTERVENTIONS:
Drug: Artesunate — 6 mg/kg/day for 2 days (total dose 12 mg/kg)
  Arms: 1
Drug: Artesunate — 4 mg/kg/day for 3 days
  Arms: 2
Drug: Mefloquine — 15mg/kg at T=0 and 10 mg/kg 6-24 hours later
  Arms: 1
Drug: Mefloquine — 8 mg/kg daily for 3 days
  Arms: 2

SUMMARY:
The main purpose of this study is to compare artesunate-mefloquine combination therapy given for 2 and 3 days at the same total dose for the treatment of uncomplicated falciparum malaria.

DETAILED DESCRIPTION:
This will be a randomized, open-label comparison of two versus three days artesunate-mefloquine treatment in patients with uncomplicated falciparum malaria. Primary endpoints will be 63-day parasitological cure rates in the 2 treatment groups. Secondary endpoints will be parasitological failure rates at each of the weekly follow-up visits to Day 56, occurence of treatment-emergent adverse events on days 0, 1 and 2, mefloquine blood concentrations on days 7, 14 and 28, and in vitro drug sensitivity profiles for parasite isolates as measured by inhibitory concentrations. Genotyping of parasites for known markers of drug resistence will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 to 70 years inclusive. If aged < 18 years the subject must have a parent or guardian in attendance.
2. Asexual stages of P. falciparum parasites in a thick or thin blood film with no other visible plasmodial species.
3. Willing to give informed consent. Parents or guardians of children and adolescents must agree to give informed consent. Assent is necessary in addition to parental informed consent.
4. Able to tolerate oral therapy.
5. Willing to attend follow-up appointments and undergo study procedures.

Exclusion Criteria:

1. History of anti-malarial drug use within the past two weeks or mefloquine (MQ) use within 4 weeks.
2. Bleeding tendency (by history or based on medical records).
3. Severe/complicated malaria as determined by the investigator (coma or seizures, pulmonary edema, shock, renal failure, jaundice, severe anemia, spontaneous bleeding, hyperparasitemia (>5% RBCs infected), or prostration).
4. History of allergy to or intolerance of study medications.
5. Mixed malaria infection by Giemsa stain.
6. Any other condition that in the opinion of the study investigator warrants parenteral antimalarial treatment.
7. Pregnant woman or nursing mother

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Determination of parasitological cure rate of directly observed antimalarial therapy | 63 days from initiation of treatment

SECONDARY OUTCOMES:
Parasitological cure rates | Weekly to Day 56
Occurence of treatment-emergent adverse events | 3 days
In vitro drug sensitivity profile for individual parasite isolates | Baseline
Mefloquine whole blood concentrations | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Wichai - Satimai, M.D., D.T.M. & H., Principal Investigator — Bureau of Vector-Borne Disease, Department of Disease Control, Ministry of Public Health; Mark M. Fukuda, M.D., Principal Investigator — Dept. of Immunology and Medicine, AFRIMS
Locations (1):
- Vector Borne Diseases Control Units (VBDC, malaria clinics), Borai, Khaosaming and Muang Districts, Changwat Trat, Thailand